CLINICAL TRIAL: NCT00243737
Title: Open-label, Stratified Study on the Efficacy, Safety and Pharmacokinetic Characteristics of Two Paediatric Formulations of ArtequinTM in Children With Acute Uncomplicated P. Falciparum Malaria
Brief Title: Efficacy, Safety and Pharmacokinetic of ArtequinTM P. Falciparum Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Schweitzer Hospital (Other)
Collaborators: Mepha Ltd. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AM-P 001-2005
Record Dates: First submitted 2005-10-24; First posted 2005-10-25 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Malaria
Keywords: Malaria; falciparum; Mefloquine; Artesunate; Artemisinin
MeSH Terms: conditions — Malaria

INTERVENTIONS:
Drug: Artesunate-Mefloquine

SUMMARY:
Treatment of Plasmodium falciparum malaria in Africa is increasingly difficult. Resistance to cheap efficient antimalarial drugs poses an increasing threat. The rapid emergence of resistance to sulfadoxine - pyrimethamine, already seen in East Africa is growing and is likely to have an striking impact on mortality in many other African regions where no obvious alternatives are available. WHO recommends the use of drug combinations containing artemisinin compounds, i.e., artemisinin-based combination therapies (ACT). Previous clinical trials have shown that the combination of artesunate with mefloquine is highly effective and well tolerated in the treatment of multidrug-resistant falciparum malaria, retaining the benefit of rapidity of action while augmenting cure rates, and apparently slowing the development of mefloquine resistance. Compliance with sequential combination regimen of antimalarial drugs is notoriously poor. Therefore, in order to limit the development of resistance to both drugs and ameliorate patients' compliance to antimalarial treatments, an optimal simultaneous combination regimen of artesunate and mefloquine in a practical single blister pack has been developed by Mepha Ltd. and successfully tested. The currently available

DETAILED DESCRIPTION:
Artequin dosages could only be tested in children able to swallow tablets and with a body weight of more than 20 kg. However, there is a great need for an Artequin formulation for smaller children unable to swallow tablets. The new Artequin Paediatric oral formulation is a flavoured, taste-masked preparation of granules of 50 mg artesunate and 125 mg mefloquine as a fixed-dose combination (once daily in one single Stickpack, i.e. 3 Stickpacks for a 3-day treatment). It is suitable for children with up to 20 kg body weight (with a range of 10-20 kg).

ELIGIBILITY:
Inclusion Criteria:

Male or female with a body weight ≥10 to 40 kg

* Patients suffering from acute uncomplicated Plasmodium falciparum malaria
* Malaria diagnosis confirmed by a positive blood smear with asexual forms of Plasmodium falciparum (i.e., identification of asexual parasite count ≥1,000 to 250,000 per mm3)
* Ear temperature 37.5°C or a history of fever within the last 48 hours
* Haemoglobin 7g/100ml
* Written informed consent and written consent from parents/guardian for children below age of consent (verbal consent in presence of literate witness is required for illiterate patients or parents/guardians).

Exclusion Criteria:

Patients with signs and symptoms of severe/complicated malaria requiring parenteral treatment (defined according to WHO Recommendations "Malaria Control Today", RBM Working Document, March 2005, see Appendix 2)

* Patients with known hypersensitivity or allergy to artemisinin derivatives or mefloquine or mefloquine chemically related compounds (for example quinine and quinidine)
* Patients who had received quinine or any artemisinin derivatives within 12 hours prior to study start
* Patients who had received any other adequate antimalarial drug therapy including antibiotics which might be active against malaria infection within 1 week prior to study start
* Patients who had received investigational (unlicensed) drugs as well as mefloquine within 30 days prior to study start
* Patients with known history of psychiatric disorders
* Patients with known history of cardiac diseases and arrhythmia
* Patients with known sickle cell disease
* Patients with clinical signs of or laboratory evidence for any other severe hepatic, renal, pulmonary, cardiac, metabolic, psychiatric, cancer or haematologic diseases
* Pregnancy or lactation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70
Dates: Start 2005-10; Study Completion 2006-04

PRIMARY OUTCOMES:
Efficacy, Proportion of patients cured on day 28

SECONDARY OUTCOMES:
Efficacy: day 14v cure rate, parasite and fever clearance time, parasite reduction rate, gametocytemia, in relation to blood concentrations of Dihydroartemisinin and mefloquine, safety, tolerability, acceptability
parasite and fever clearance time, parasite reduction rate, gametocytemia, in relation to blood concentrations of Dihydroartemisinin
  Time to complete clearance of fever and parasitemia Assessment in relation to DHA and mefloquine blood levels
safety, tolerability, acceptability
  Assessment of adverse events and reporting of tolerability, safety and acceptability

CONTACTS AND LOCATIONS:
Overall Officials: Maryvonne Kombila, Prof Dr, Principal Investigator — Département de Parasitologie-Mycologie, Faculté de médecine
Locations (2):
- Gabon (2):
  - Medical Research Unit, Albert Schweitzer Hospital, Lambaréné
  - Département de Parasitologie-Mycologie, Faculte de medecine, Libreville

REFERENCES:
- [Derived] Bouyou-Akotet MK, Ramharter M, Ngoungou EB, Mamfoumbi MM, Mihindou MP, Missinou MA, Kurth F, Belard S, Agnandji ST, Issifou S, Heidecker JL, Trapp S, Kremsner PG, Kombila M. Efficacy and safety of a new pediatric artesunate-mefloquine drug formulation for the treatment of uncomplicated falciparum malaria in Gabon. Wien Klin Wochenschr. 2010 Mar;122(5-6):173-8. doi: 10.1007/s00508-010-1317-1. PMID 20361381